CLINICAL TRIAL: NCT03031951
Title: Lifestyle Intervention Program for Former Elite Athletes
Acronym: Champ4Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Motricidade Humana (Other)
Responsible Party: Principal Investigator, Analiza Mónica Lopes Almeida Silva, Assistant Professor, Faculdade de Motricidade Humana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 16/2016
Record Dates: First submitted 2017-01-16; First posted 2017-01-26 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Obesity
Keywords: Former athletes; Body composition; Adaptive thermogenesis; Physical activity; Energy expenditure; Sedentary behavior; Fat mass; Abdominal fat mass; Nutrition; Behavior modification
MeSH Terms: conditions — Obesity; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle Intervention Group (Experimental): Subjects will attend 12 educational sessions for a healthy lifestyle in groups of 10-15 participants, for approximately 4 months. Sessions will last 90-120 minutes and will include educational content and practical application classroom exercises in the areas of physical activity and exercise, diet and eating behavior, and behavior modification. The inclusion of self-regulation skills, such as pedometer use, recording food regularly and monitoring weight, is also part of the curriculum. Participants will be instructed and motivated to make small but enduring reductions in caloric intake and to increase energy expenditure to induce a daily energy deficit of approximately 300 kcal. Weight will be monitored weekly.
  Interventions: Behavioral: Lifestyle Intervention Group
- Control Group - Waiting List (No Intervention): Participants assigned to the control group will have access to the intervention after the 12-month period - waiting list. Meanwhile, participants will receive multimedia health information fortnightly by e-mail over the first 4-month period. The health information covers healthy lifestyle topics.
  During the 12 months of study participation, control group participants will be instructed to maintain their baseline level of physical activity. Individuals assigned to the control group will be asked to maintain their current nutritional practices and physical activity patterns.

INTERVENTIONS:
Behavioral: Lifestyle Intervention Group — The intervention group will start the lifestyle intervention with a 60-minute nutrition appointment given by a certified dietitian. This meeting is intended to provide a well-balanced personalized diet plan, calculated to create a moderate reduction from ~300 to 500kcal/day according to each participant's energy requirements and preferences. Two additional follow-up appointments are also planned to adjust the individual energy requirements throughout the intervention. Subjects will attend 12 educational sessions for a healthy lifestyle in groups of 10-15 participants, for approximately 4 months. Sessions will last 60-90 minutes and will include educational content and practical application classroom exercises in the areas of physical activity and exercise, diet and eating behavior, and behavior modification. The inclusion of self-regulation skills, such as pedometer use, recording food regularly and monitoring weight, is also part of the curriculum. Weight will be monitored weekly.
  Other Names: Lifestyle Intervention Programme
  Arms: Lifestyle Intervention Group

SUMMARY:
Given the lack of support for lifestyle management in post-career and considering the high rates of physical inactivity and overweight in former elite athletes, the aim of this research project is to analyze the efficacy and effectiveness of a lifestyle intervention in former athletes.

DETAILED DESCRIPTION:
The physical preparation of the elite athlete results from a complex and very demanding daily training. In this process high energy expenditure (EE) occur compensated by a proportional energy intake, thus contributing to neutral energy balance and weight maintenance. However, a positive energy balance (and consequently an increase in weight) is expected after the end of the sports career if the energy intake is maintained for lower EE. While clinicians and researchers are concerned with the average individual whose physical activity (PA) level is far below the recommended exercise dose an often overlooked group are the former highly competitive athletes, who have been exposed to higher amounts of vigorous PA during times of training and competition.

It is common that upon retirement energy intake does not match the dramatic decrease in overall energy expenditure leading to a positive energy balance, and consequently weight gain. The change to a lower physical activity level does not induce an equivalent reduction in energy intake. Varying physical activity level from 1.8 to 1.4 over 7 days was not associated with a change of energy intake and there was no tendency for energy intake to drop as the sedentariness progressed.

In fact, elite athletes that became inactive are susceptible to various chronic diseases such as obesity, diabetes and cardiovascular disease. Not only obesity and its comorbidities are a major health problem as an increase in body weight and a higher risk for developing hypertension, type II diabetes and cardiovascular disease has been observed in athletes that retired from the sports career . However, the literature reports that this risk is only present in those retired athletes exposed to a sedentary lifestyle. In fact, the current levels of PA are more protective against the development of cardiovascular disease in former athletes than their past sports history. Although it is expected that the retired elite athlete will be engaged in regular PA throughout life, studies reveal that this assumption does not apply to all former athletes. This concern was addressed in the United States, namely within the National Football League where an obesity prevention program for the retired athletes was implemented. In Portugal ~50% of the former elite athletes are overweight/obese and ~30% are inactive, based on self-reports measures. Indeed no support is provided for maintaining a healthy lifestyle after the end of the sports career. If a healthy lifestyle promotion among post-career elite athletes would contribute to avoid the observed rates of overweight/obesity it is unknown. Considering this actual context, the aim of this research project is to analyze the effect of a lifestyle intervention in former athletes. To accomplish the goals the investigators will perform a 1 year randomized controlled trial with a 4-month lifestyle intervention and an 8-month follow-up in 100 volunteered former overweight (Body Mass index>25 kg.m-2), inactive elite athletes that represented Portugal in international competitions during 1972-2012, ended their career for at least 2 years prior the study and are able to attend the educational sessions. Participants will be randomly assigned into 2 groups: i) dietary counseling (control group), or ii) behavioral lifestyle intervention, focusing on diet and PA. All participants will be screened at baseline, 4 months, and 12 months. A broad set of parameters will be assayed in each participant, namely: body composition, cardiorespiratory fitness, muscle strength, biochemical parameters, resting metabolic rate, nutritional intake, daily PA, and quality of life. These variables will allow the comprehension of the effects of a lifestyle modification on fatness, fitness and health-related parameters contributing also to further elucidate compensatory mechanisms associated with potential changes in weight and composition. To accomplish the main goal the research team will use established methods in the literature as well as novel procedures, which will enable the research team to overcome some of the limitations of previous studies. At the end of the study the investigators expect to have collected consistent data about whether a lifestyle intervention is or is not able to effectively decrease fatness while improving fitness and health-related markers. The research team believe that these data will help both non-governmental and governmental stakeholders in sports and education to make evidence based decisions, specifically the introduction and implementation of lifestyle programs in the transition to the post-career of elite athletes. The growing number of elite athletes supported by the government along with the recent EU report guidelines on dual careers in high-performance sports (ec.europa.eu/sport/news/2013/20130123-eu-guidelines-dualcareers_en.htm) requires further studies that test the role of preventive and educational programs for athletes in the areas of healthy living. The past experience of the research team in body composition, physical fitness, and objectively measured PA using cross-sectional and prospective study designs in athletic and non-athletic populations, as well as in the conduction of PA intervention clinical trials, together with the involvement of the Portuguese Olympic Committee as partners, supports the chances of successfully achieving the proposed objectives.

ELIGIBILITY:
Inclusion Criteria:

* Being a Former high-level athlete;
* Being Physical Inactive (not exercising for >20 min at least 3 days/week);
* Being Overweight or Obese (BMI exceed≥25 kg/m2);
* Willing to be randomized to either control or intervention groups and follow the protocol to which they have been assigned;
* Willing to participate in the educational sessions performed at Faculdade de Motricidade Humana - Universidade de Lisboa;
* Unwilling to consider using weight loss medications;

Exclusion Criteria:

* Failure to complete the run-in for dietary intake and physical activity;
* Lack of support from primary health care provider or family members;
* Being unable or unwilling to give informed consent or communicate with local study staff;
* Current diagnosis of schizophrenia, other psychotic disorders, or bipolar disorder;
* Eating disorders;
* Medical conditions such as thyroid disorders;
* Diabetes and cardiovascular disease or other medical condition known to affect energy balance homeostasis;
* Hospitalization for depression in past six months;
* Self-report of alcohol or substance abuse within the past twelve months, current consumption of more than 14 alcoholic drinks per week, and/or current acute treatment or rehabilitation program for these problems;
* Pregnancy or planning to get pregnant within the next 9 month, having been pregnant within the past 6 months or breastfeeding;
* History of weight loss surgery or liposuction procedures;
* Current participation in a weight loss program;
* In the past three months, weight loss exceeding 4.5 kg (such individuals may have difficulty losing additional weight) or successful attempts to lose weight within the past 6-month;
* Current use of medications for weight loss;
* Chronic treatment with systemic corticosteroids;
* Self-reported inability to walk two blocks;
* Inability to complete the study within the designated time frame because of plans to move out of the study area;
* Inability to attend the visits/appointments, evaluation measurements, and attend the intervention sessions at the Faculdade de Motricidade Humana - Universidade de Lisboa;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2016-09; Primary Completion 2020-10 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Whole body fat mass (FM) | 12 month
  To estimate total FM, dual energy X-ray absorptiometry (Hologic Explorer-W, Waltham, USA) will be used. A whole-body scan will be performed and the attenuation of X-rays pulsed between 70 and 140 kV synchronously with the line frequency for each pixel of the scanned image will be measured.
  Total abdominal FM by identifying a specific region of interest (ROI) within the analysis programme.
Abdominal Fat Mass | 12 months
  Specific DXA ROIs for abdominal regional fat will be defined as follows: ROI 1, the upper edge of the second lumbar vertebra (approximately 10 cm above the L4 to L5) to above the iliac crest and laterally encompasses the entire breadth of the abdomen, thus determining total abdominal fat mass.

SECONDARY OUTCOMES:
Weight | 12 months
  Subjects will have their weight measured (in kilograms) wearing a bathing suit to the nearest 0.01 kg with a weight scale (Seca, Hamburg, Germany)
Height | baseline
  Subjects will have their height measured (in meters) without shoes to the nearest 0.1 cm with a stadiometer (Seca, Hamburg, Germany).
Body mass index | 12 months
  Weight (in kilograms) and height (in meters) will be combined to report BMI in kg/m^2.
Circumferences | 12 months
  Subjects will have their. Waist circumference will be measured immediately above the iliac crest. Hip circumference will be assessed is determined at the maximum perimeter of the hips. Arm and thigh circumferences will be assessed at the level of the skinfold measurement. Calf circumference will be assessed at the at the maximum perimeter of the calf. Circumference measurements are performed twice and the arithmetic mean of both values is considered as the final value.
Cardiorespiratory Fitness | 12 months
  Maximal oxygen uptake (VO2max) capacity will be assessed using the Bruce maximal exercise test protocol performed on a variable speed and incline treadmill (Quinton Treadmill, Model 640, 90TM Series). VO2max is achieved when at least 2 of the following 3 criteria are obtained: a heart rate at or above the age-predicted maximum, and/or a respiratory exchange ratio greater than 1, and/or no increase in VO2max despite further grade increases.
Systolic blood pressure | 12 months
  Three measurements of systolic blood pressure are obtained with the participant in the sitting position using a digital sphygmomanometer. The blood pressure cuff-fixed on the nondominant upper arm is loosened during the two minutes pause between the measurements. The arithmetic means of the second and third reading are considered as the participants' blood pressure and pulse values, respectively. Overall, there is a rest of approximately five minutes before the second blood pressure measurement is carried out
Diastolic blood pressure | 9 months
  Three measurements of diastolic blood pressure are obtained with the participant in the sitting position using a digital sphygmomanometer. The blood pressure cuff-fixed on the nondominant upper arm is loosened during the two minutes pause between the measurements. The arithmetic means of the second and third reading are considered as the participants' blood pressure. Overall, there is a rest of approximately five minutes before the second blood pressure measurement is carried out
Blood Glucose levels | 12 months
  Blood glucose levels will be performed in serum samples using coloured enzymatic tests, in an automated analyser (Cobas Integra 400).
Blood lipid profiles | 12 months
  Blood lipid profile, including total cholesterol, high density lipoprotein cholesterol (HDL) will be performed in serum samples using coloured enzymatic tests, in an automated analyser (Cobas Integra 400).
Blood insulin levels | 12 months
  Blood insulin levels assessment will be performed in an automated analyser (Cobas Integra 400) by eletroquimioluminescence.
Blood thyroid levels | 12 months
  Blood thyroid panel (T3, T4, TSH) will be run by immunoassay with chemiluminescent detection (Millipore Corp., Billerica, MA).
Blood leptin levels | 12 months
  Serum levels of leptin will be measured by ELISA.
Lower muscle strength | 12 months
  One repetition leg press maximum test (1RM) that measure the maximal weight a subject can lift with one repetition will be used. Before each assessment the participant will be instructed to conduct a 5min warmup period, preceded by a respective familiarization period with the specific test for the lower limb. The evaluation of the maximum strength of the leg will be made by performing a horizontal leg press isometric test (S0409, BPH) with the bent leg and the knee joint at an angle of 110 °. Participants will complete 5 maximal voluntary repetitions lasting 34 seconds, and a period of rest between reps 60s. All participants will be asked to produce strength the fastest possible in all repetitions. The Plux software (Biosignalsplux) will be considered to analyze the highest value between the maximal voluntary repetitions.
Upper muscular strength | 12 months
  Handgrip strength test evaluates maximal isometric force of the forearm muscle and will be assessed by a portable hand dynamometer JAMAR plus digital (Sammons Preston, Bolingbrook, IL). Participants will be assessed on both hands alternately. Prior to the test, the grip dynamometer will be adjusted to the size of the hand of each subject. Each participant will be assessed on both hands alternately until add up three attempts for each hand. In each attempt the subject will exert the maximal grip strength on the handgrip dynamometer with the assessed hand during 5 seconds. After each attempt there will be a resting period of 60 seconds that will be used both for recovery and for changing the handgrip dynamometer to the opposite hand.
Eating self-regulation markers | 12 months
  The reward value of food (i.e., implicit wanting/explicit liking and wanting) will be measured by a computer procedure, the Leeds Food Preference Questionnaire (LFPQ) [38, 39], which uses a 'forced choice' reaction time measure of implicit wanting in addition to explicit subjective measures of liking and wanting for visual food stimuli varying in fat content and taste. Implicit wanting is operationalized as the reaction time of each pair trial decision. Thus, the speed with which one category of stimuli is chosen relative to alternative categories provides a quantifiable measure of implicit wanting for each food category in the procedure.
Exercise Motivation | 12 months
  The Behavioral Regulation in Exercise Questionnaire - 3 (BREQ-3) will be used to assess motivations to engage in exercise. BREQ-3 contains 24 items, organized into 6 subscales, measuring amotivation, external, introjected (i.e controlled motivational regulations), identified, integrated, and intrinsic motivations (i.e autonomous motivational regulations). Following the stem "why do you exercise", participants respond on a 5-point Likert scale ranging from 0 ("not true for me") to 4 ("very true for me"). Prior research has supported BREQ's factor structure and reliability (Cronbach's alphas > 0.70).
Raw BIA parameters - Resistance and Reactance | 12 months
  Whole body R (Ω) and Xc (Ω) will be assessed by Bioelectrical impedance spectroscopy analysis (model 4200B; Xitron Technologies, San Diego, CA, USA) and by a single-frequency BIA, phase-sensitive 50 kHz (BIA-101, RJL/Akern Systems, Firenze, Italy).
  Before the test, subjects were instructed to lie in a supine position with their arms and legs abducted at a 458 angle for 10 min. This impedance spectra was modelled with the Cole-Cole cell suspension model to derive a theoretical impedance at zero and infinity frequency, based on a non-linear curve fitting from the measured resistance and reactance.
Raw BIA parameters - Phase Angle | 12 months
  Phase angle (º) will be assessed by Bioelectrical impedance spectroscopy analysis (model 4200B; Xitron Technologies, San Diego, CA, USA). Before the test, subjects were instructed to lie in a supine position with their arms and legs abducted at a 458 angle for 10 min. This impedance spectra was modelled with the Cole-Cole cell suspension model to derive a theoretical impedance at zero and infinity frequency, based on a non-linear curve fitting from the measured resistance and reactance. The frequency 50 kHz will be used for phase angle analysis.
Total body water, Intracellular water and Extracellular water | 12 months
  Intracellular water and extracellular water were predicted from the Hanai mixture theory, and TBW was estimated by the sum of intracellular water and extracellular water. Considering ten repeated measures, the TEM and CV for TBW were 0·47 litres and 1·1% respectively.
Macronutrient composition of the diet | 12 months
  Food records will also be collected to characterize macronutrient composition of the diet in the 3 moments using a software package (Food Processor SQL, ESHA Research, Salem, OR, USA).
Energy Intake | 12 months
  When total energy expenditure (TEE) is obtained in conjunction with measured body composition, then two terms of the energy balance equation are known, namely ES and EE. From equation 1 it is possible to solve for average energy intake during the course of the study.
  The magnitude of compensation will be calculated as the difference between achieved energy imbalance and energy expenditure.
Free-living physical activity | 12 months
  The amount of activity assessed by the Actigraph accelerometer will be expressed as minutes per day spent in different intensities. The cutoff values used to define the intensity of PA and therefore to quantify the mean time in each intensity (sedentary, light, moderate or vigorous) will be: sedentary: < 100 counts·min-1; light: 100-2019 counts·min-1; moderate: 2020-5998 counts·min-1 (corresponding to 3-5.9 METs); vigorous: ≥ 5999 counts·min-1 (corresponding to ≥6 METs). The Actiheart (Actiheart, CamNtech Limited, UK) is a lightweight (10 g) combined heart rate (HR) and movement (uniaxial accelerometer oriented to measure acceleration along the body's longitudinal axis) sensor that utilizes both piezoelectric accelerometer and HR data synchronously. Participants will wear the Actiheart 24h day-1 at the same time as the accelerometer and a valid day will be defined as having 600 or more minutes (≥10h) of monitor wear during waking hours.
Total energy expenditure | 12 months
  Total energy expenditure will be assessed by the Actigraph accelerometer using the Crouter et al equations.
Physical activity energy expenditure | 12 months
  Physical activity energy expenditure (PAEE) will be calculated as total energy expenditure (TEE) minus (0.1*TEE + REE), assuming the termic effect of food represents 10% of TEE, and REE represents Resting energy expenditure.
Adaptive Thermogenesis | 3 and 9 months
  In order to predict resting energy expenditure (REE) at baseline, a gender specific regression equation using FFM and FM as the independent predictor will be generated. This equation will then be used to predict REE at 3 and after a 9-month follow-up, using the measured values of FM and FFM at these time points. To disclose any adaptations in REE not accounted for by changes in FFM, adaptive response will be assessed as 1 minus the ratio between the actual to the expected/predicted REE, multiplied by 100. Positive values indicate a decrease in REE beyond that expected by changes in body composition (actual REE below predicted REE) whereas negative values represent a change in REE equal to or greater than the predicted REE (actual REE higher than predicted REE).
Resting Energy Expenditure (REE) | 12 months
  The MedGraphics CPX Ultima (MedGraphics Corporation, Breezeex Software) indirect calorimeter will be used to measure breath-by-breath oxygen consumption (V̇O2 ) and carbon dioxide production (V̇CO2) using a facial mask. The oxygen and carbon dioxide analyzers will be calibrated in the morning before testing using known gas concentration. Before testing, participants will be instructed about all the procedures and asked to relax, breathe normally, not to sleep, and not to talk during the evaluation. Total rest duration will be 45 minutes, participants lied supine for 15 minutes covered with a blanket and the calorimeter device will then be attached to the mask and breath by breath V̇O2 and V̇CO2 will be measured for 30 min period.
  The mean V̇O2 and V̇CO2 of 5 min steady states will be used in Weir equation and the period with the lowest REE will be considered for data analysis.
Reported Quality of Life | 12 months
  To measure general health-related quality of life, participants will complete the Short-Form Health Survey (SF-36) questionnaire [45], with a total of 36 items composed of eight dimensions: Physical functioning (Cronbach's a = .83), physical role limitations (Cronbach's a = .89), bodily pain (Cronbach's a = .88), general health (Cronbach's a = .82), emotional role limitations (Cronbach's a = .74), social functioning (Cronbach's a = .71), vitality (Cronbach's a = .86), and mental health (Cronbach's a = .90). Higher scores indicate better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Analiza Silva, Principal Investigator — Faculty of Human Kinetics, University of Lisbon
Locations (1):
- Faculdade de Motricidade Humana, Oeiras, Cruz-Quebrada, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stubbs RJ, Hughes DA, Johnstone AM, Horgan GW, King N, Blundell JE. A decrease in physical activity affects appetite, energy, and nutrient balance in lean men feeding ad libitum. Am J Clin Nutr. 2004 Jan;79(1):62-9. doi: 10.1093/ajcn/79.1.62. PMID 14684398
- [Background] Miller MA, Croft LB, Belanger AR, Romero-Corral A, Somers VK, Roberts AJ, Goldman ME. Prevalence of metabolic syndrome in retired National Football League players. Am J Cardiol. 2008 May 1;101(9):1281-4. doi: 10.1016/j.amjcard.2007.12.029. Epub 2008 Mar 7. PMID 18435958
- [Background] Pihl E, Jurimae T. Relationships between body weight change and cardiovascular disease risk factors in male former athletes. Int J Obes Relat Metab Disord. 2001 Jul;25(7):1057-62. doi: 10.1038/sj.ijo.0801642. PMID 11443506
- [Background] Pihl E, Zilmer K, Kullisaar T, Kairane C, Magi A, Zilmer M. Atherogenic inflammatory and oxidative stress markers in relation to overweight values in male former athletes. Int J Obes (Lond). 2006 Jan;30(1):141-6. doi: 10.1038/sj.ijo.0803068. PMID 16158088
- [Background] Dey SK, Ghosh C, Debray P, Chatterjee M. Coronary artery disease risk factors & their association with physical activity in older athletes. J Cardiovasc Risk. 2002 Dec;9(6):383-92. doi: 10.1097/01.hjr.0000049244.21319.20. PMID 12478209
- [Background] Kujala UM, Marti P, Kaprio J, Hernelahti M, Tikkanen H, Sarna S. Occurrence of chronic disease in former top-level athletes. Predominance of benefits, risks or selection effects? Sports Med. 2003;33(8):553-61. doi: 10.2165/00007256-200333080-00001. PMID 12797837
- [Background] Buchwald H, Roberts AJ. The HOPE (heart, obesity, prevention, education) program for former NFL players. Surg Obes Relat Dis. 2014 Jul-Aug;10(4):573-5. doi: 10.1016/j.soard.2014.02.030. Epub 2014 Mar 1. No abstract available. PMID 24958646
- [Background] Batista C, Soares JM. Are former athletes more prone to asthma? J Asthma. 2013 May;50(4):403-9. doi: 10.3109/02770903.2013.776075. Epub 2013 Apr 8. PMID 23489224
- [Derived] Nunes CL, Jesus F, Rosa GB, Marianito M, Francisco R, Bosy-Westphal A, Minderico CS, Martins P, Sardinha LB, Silva AM. Interindividual variability in energy intake and expenditure during a weight loss intervention. Appetite. 2024 Feb 1;193:107162. doi: 10.1016/j.appet.2023.107162. Epub 2023 Dec 13. PMID 38101517
- [Derived] Nunes CL, Rosa GB, Jesus F, Heymsfield SB, Minderico CS, Martins P, Sardinha LB, Silva AM. Interindividual variability in metabolic adaptation of non-exercise activity thermogenesis after a 1-year weight loss intervention in former elite athletes. Eur J Sport Sci. 2023 Aug;23(8):1761-1770. doi: 10.1080/17461391.2022.2147020. Epub 2022 Nov 28. PMID 36377398
- [Derived] Nunes CL, Carraca EV, Jesus F, Finlayson G, Francisco R, Silva MN, Santos I, Bosy-Westphal A, Martins P, Minderico C, Sardinha LB, Silva AM. Changes in food reward and intuitive eating after weight loss and maintenance in former athletes with overweight or obesity. Obesity (Silver Spring). 2022 May;30(5):1004-1014. doi: 10.1002/oby.23407. Epub 2022 Mar 28. PMID 35347875
- [Derived] Nunes CL, Jesus F, Francisco R, Matias CN, Heo M, Heymsfield SB, Bosy-Westphal A, Sardinha LB, Martins P, Minderico CS, Silva AM. Adaptive thermogenesis after moderate weight loss: magnitude and methodological issues. Eur J Nutr. 2022 Apr;61(3):1405-1416. doi: 10.1007/s00394-021-02742-6. Epub 2021 Nov 27. PMID 34839398
- [Derived] Silva AM, Nunes CL, Jesus F, Francisco R, Matias CN, Cardoso M, Santos I, Carraca EV, Finlayson G, Silva MN, Dickinson S, Allison D, Minderico CS, Martins P, Sardinha LB. Effectiveness of a lifestyle weight-loss intervention targeting inactive former elite athletes: the Champ4Life randomised controlled trial. Br J Sports Med. 2022 Apr;56(7):394-401. doi: 10.1136/bjsports-2021-104212. Epub 2021 Oct 1. PMID 34598935
- [Derived] Matias CN, Campa F, Nunes CL, Francisco R, Jesus F, Cardoso M, Valamatos MJ, Homens PM, Sardinha LB, Martins P, Minderico C, Silva AM. Phase Angle Is a Marker of Muscle Quantity and Strength in Overweight/Obese Former Athletes. Int J Environ Res Public Health. 2021 Jun 21;18(12):6649. doi: 10.3390/ijerph18126649. PMID 34205575
- [Derived] Campa F, Matias CN, Nunes CL, Monteiro CP, Francisco R, Jesus F, Marini E, Sardinha LB, Martins P, Minderico C, Silva AM. Specific Bioelectrical Impedance Vector Analysis Identifies Body Fat Reduction after a Lifestyle Intervention in Former Elite Athletes. Biology (Basel). 2021 Jun 12;10(6):524. doi: 10.3390/biology10060524. PMID 34204604